CLINICAL TRIAL: NCT00067197
Title: Modulation of Motor Learning in Chronic Stroke Patients by Transcranial DC Stimulation
Brief Title: Improving Motor Learning in Stroke Patients
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030267; 03-N-0267
Record Dates: First submitted 2003-08-12; First posted 2003-08-13 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-07-17

CONDITIONS: Cerebrovascular Accident
Keywords: Transcranial Direct Current Stimulation (tDCS); Cortical Reorganization; Rehabilitation; Motor Learning; Activity of Daily Living (ADL); Stroke; Healthy Volunteer; HV
MeSH Terms: conditions — Stroke

SUMMARY:
No universally successful therapy exists that promotes recovery of motor function after a stroke, the main cause of long-term disability among adults.

The purpose of this study is to develop strategies to improve recovery of lost motor function. It will combine motor skills training with a brain-stimulating technique called transcranial direct current stimulation (tDCS).

Healthy adult volunteers and adult stroke patients will be enrolled in this study. Participants will come to NIH for a clinical and neurological exam, and, if necessary, an MRI [magnetic resonance imaging] examination. Participants will return for 4 sessions; each lasting approximately 3 hours. The first will be a practice session during which participants will become familiar with the motor skills required of them in this study, such as performing finger movements on a keyboard, pinching, tapping, making wrist movements, and lifting small items. In sessions 2 and 3, participants will perform the motor skills they practiced in session 1 while receiving tDCS. During session 4, they will receive tDCS only, with no performance of motor skills.

During tDCS, investigators will place electrodes with a gel on participants' heads and pass the tDCS current between these two electrodes. tDCS is a painless procedure.

Participants will receive up to $420 in compensation for their involvement in this study.

...

DETAILED DESCRIPTION:
There is no universally accepted strategy to promote recovery of motor function after chronic stroke, the main cause of long-term disability among adults. It is desirable to develop strategies to accelerate motor learning in this patient group. Previous studies in healthy volunteers demonstrated that cortical stimulation in association with training leads to improvements of motor learning and use-dependent plasticity. The purpose of this protocol is to apply a painless stimulation technique to the motor cortex of the affected hemisphere of patients with subcortical stroke (transcranial DC stimulation, tDCS) to test the hypothesis that tDCS of the motor cortex of the affected hemisphere in association with motor training will improve motor learning of a finger sequence in the paretic hand.

Furthermore, recent studies have demonstrated that the unaffected hemisphere exerts abnormally high inhibitory influence over the affected hemisphere. This abnormality might adversely influence motor recovery. Therefore a further purpose of the study is to apply tDCS to the unaffected hemisphere to test the hypothesis that reduction of the inhibitory influence of the unaffected hemisphere over the affected in association with motor training will improve motor learning.

This technique has been so far applied in several hundred subjects worldwide in the absence of undesirable side effects reported to date.

We plan to study patients with chronic strokes and healthy age- and gender matched normal volunteers. Primary outcome measure will be the number of correct keyboard piano sequences played in a specific time-period (30 seconds). Secondary outcome measures are speed of tapping with only one finger; simple reaction times; pinch force; and a functional measure of activities of daily life (ADL): Jebsen-Tailor-Test. To better understand the mechanisms underlying the proposed behavioral gains, we will use TMS to identify changes in corticomotor excitability.

ELIGIBILITY:
* INCLUSION CRITERIA:

We will include patients with thromboembolic non-hemorrhagic hemispheric lesions at least 3 months after the stroke.

We will choose Patients who initially had a severe motor paresis (below MRC grade 2), which subsequently recovered to the point that they have a residual motor deficit but can perform the required tasks. Assessment of the initial functional state will be taken either from patient report or medical records.

As the control group, we will include age- and gender matched Normal Volunteers with matched non-dominant/dominant hand (to the affected hand of the stroke patients).

EXCLUSION CRITERIA:

Patients with more than one stroke in the medical cerebral artery territory.

Patients with bilateral motor impairment.

Patients with cerebellar or brainstem lesions.

Patients or Normal Volunteers unable to perform the task (wrist or elbow flexion at least MRC grade 2).

Patients or Normal Volunteers with severe alcohol or drug abuse, psychiatric illness like severe depression, poor motivational capacity, or severe language disturbances, particularly of receptive nature or with serious cognitive deficits (defined as equivalent to a mini-mental state exam score of 23 or less).

Patients or Normal Volunteers with history of severe uncontrolled medical problems (e.g. cardiovascular disease, severe rheumatoid arthritis, active joint deformity of arthritic origin, active cancer or renal disease, any kind of end-stage pulmonary or cardiovascular disease, or a deteriorated condition due to age, uncontrolled epilepsy or others).

Patients or Normal Volunteers with increased intracranial pressure as evaluated by clinical means.

Patients or Normal Volunteers with unstable cardiac arrhythmia.

Patients or Normal Volunteers with h/o hyperthyroidism or individuals receiving drugs acting primarily on the central nervous system.

Patients and Normal Volunteers with more than moderate to severe microangiopathy, polyneuropathy, diabetes mellitus, or ischemic peripheral disease.

Patients or Normal Volunteers which are or which have been professional piano players.

Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76
Dates: Start 2003-08-11; Study Completion 2008-07-17

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Nitsche MA, Paulus W. Sustained excitability elevations induced by transcranial DC motor cortex stimulation in humans. Neurology. 2001 Nov 27;57(10):1899-901. doi: 10.1212/wnl.57.10.1899. PMID 11723286
- [Background] Nitsche MA, Paulus W. Excitability changes induced in the human motor cortex by weak transcranial direct current stimulation. J Physiol. 2000 Sep 15;527 Pt 3(Pt 3):633-9. doi: 10.1111/j.1469-7793.2000.t01-1-00633.x. PMID 10990547
- [Background] Karni A, Meyer G, Jezzard P, Adams MM, Turner R, Ungerleider LG. Functional MRI evidence for adult motor cortex plasticity during motor skill learning. Nature. 1995 Sep 14;377(6545):155-8. doi: 10.1038/377155a0. PMID 7675082